CLINICAL TRIAL: NCT07263217
Title: Mechanistic Study on the Protective and Regenerative Effects of Spirulina in Hepatectomy-Related Liver Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0805
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — maltodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina treatment group (Experimental): participants take spirulina tablets (2 g/day) for 3 weeks before and 3 weeks after surgery.
  Interventions: Dietary Supplement: Spirulina
- Placebo control group (Placebo Comparator): participants take placebo tablets (maltodextrin, same dosage and schedule).
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Spirulina — participants take spirulina tablets (2 g/day) for 3 weeks before and 3 weeks after surgery
  Arms: Spirulina treatment group
Dietary Supplement: Maltodextrin — Participants take placebo tablets (maltodextrin, same dosage and schedule).
  Arms: Placebo control group

SUMMARY:
The goal of this clinical trial is to learn if spirulina can help protect the liver and promote recovery after partial hepatectomy (surgery to remove part of the liver). It will also learn about the safety of spirulina in patients undergoing liver surgery.

The main questions it aims to answer are:

Does spirulina help improve liver function after surgery? Does spirulina promote liver regeneration and reduce inflammation? What side effects, if any, occur when participants take spirulina? Researchers will compare spirulina tablets to a placebo (a look-alike tablet that contains no spirulina) to see if spirulina helps protect the liver and support recovery after surgery.

Participants will:

Take spirulina or placebo tablets daily for 3 weeks before and 3 weeks after surgery.

Provide blood and stool samples before and after treatment. Allow the collection of a small piece of liver tissue (from surgical waste) for analysis.

Have regular clinic visits for checkups, blood tests, and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cholangiocarcinoma (bile duct cell carcinoma).
* Child-Pugh Class A liver function.
* Planned to receive neoadjuvant therapy with gemcitabine + oxaliplatin, combined with lenvatinib and a PD-1 inhibitor, followed by anatomical hemihepatectomy (remaining liver volume > 40%).
* Age 18-75 years, male or female. Willing and able to comply with the study protocol, including oral administration of spirulina or placebo for 3 weeks before and 3 weeks after surgery.
* Voluntarily agrees to participate and signs written informed consent.
* Has had no acute illness or significant symptom worsening within 4 weeks before enrollment.

Exclusion Criteria:

* Presence of severe comorbidities (e.g., uncontrolled cardiovascular, respiratory, renal, or hematologic diseases).
* Known allergy to spirulina or its components.
* Concurrent malignant tumors other than the target disease.
* History of previous liver resection surgery.
* Severe psychiatric disorders that could affect compliance or the ability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Alanine Aminotransferase (ALT) Level | Day 0 (pre-treatment, ~3 weeks before surgery) End of 6-week treatment (~3 weeks after surgery)
  Serum ALT will be measured at baseline and after the 6-week perioperative intervention. The outcome is the change from baseline compared between spirulina and placebo groups.
Change in Aspartate Aminotransferase (AST) Level | Day 0 (~3 weeks before surgery) End of 6-week treatment (~3 weeks after surgery)
  Serum AST will be measured at baseline and after the intervention. The analysis compares change from baseline between study arms.
Change in Total Bilirubin (TBIL) Level | Day 0 (~3 weeks before surgery) End of 6-week treatment (~3 weeks after surgery)
  Serum TBIL will be measured pre- and post-intervention. The change from baseline will be compared between groups.

SECONDARY OUTCOMES:
Change in Serum Inflammatory Cytokine Concentrations | Day 0 (~3 weeks before surgery) End of 6-week treatment (~3 weeks after surgery)
  Serum inflammatory cytokines (e.g., IL-6, TNF-α) will be quantified using immunoassays before and after intervention. Analysis will compare changes from baseline.
Change in Gut Microbial Species Abundance Measured by Fecal Metagenomic Sequencing | Day 0 (~3 weeks before surgery) End of 6-week treatment (~3 weeks after surgery)
  Fecal metagenomic sequencing will assess gut microbial species abundance and alpha-diversity indices. The outcome is change in microbial composition from baseline to post-treatment.
Gene Expression Profiles from Liver Tissue Assessed by Single-cell and/or Bulk Transcriptomic Sequencing | During liver surgery (partial hepatectomy)
  Single-cell RNA sequencing and/or bulk RNA sequencing will be performed on liver tissue collected during partial hepatectomy to characterize cellular and molecular pathways related to liver injury and regeneration.

OTHER OUTCOMES:
Number of Participants With Abnormal Hematology Laboratory Values | Day 0 (baseline) Perioperative period (during hospitalization) End of 6-week treatment (~3 weeks after surgery)
  Complete blood count parameters will be assessed at baseline, during intervention, and at end of treatment. The outcome is the number of participants exhibiting abnormal values defined by institutional reference ranges.
Number of Participants With Abnormal Renal Function Test Results | Day 0 Perioperative period End of 6-week treatment
  Renal function parameters including serum creatinine and blood urea nitrogen will be assessed. The number of participants with abnormal values will be reported.
Number of Participants With Abnormal Coagulation Function Test Results | Day 0 Perioperative period End of 6-week treatment
  Coagulation parameters including prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (APTT) will be collected. Abnormal findings will be counted.
Number of Participants With Abnormal Urine Routine Test Results | Day 0 Perioperative period End of 6-week treatment
  Routine urinalysis including leukocytes, nitrites, protein, glucose, ketones, and microscopic examination will be performed. Abnormal results will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, China